CLINICAL TRIAL: NCT03724331
Title: Understanding the Post-Surgical Non-Small Cell Lung Cancer Patient's Symptom Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Corewell Health West (Other); National Cancer Institute (NCI) (NIH); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0560-18-EP; R01CA205025 (NIH)
Record Dates: First submitted 2018-10-25; First posted 2018-10-30 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Fatigue; Self Efficacy; Quality of Life; Physical Activity; Lung Cancer; Non-Small Cell Lung Cancer
Keywords: Cancer-Related Fatigue; Fatigue; Symptoms; Functional Status; Quality of Life; Lung Cancer; Rehabilitation; Exercise; Physical Activity; Self-Efficacy; Self-Management
MeSH Terms: conditions — Fatigue; Motor Activity; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Light Physical Activity 1 (Experimental): Conventional treatment for cancer as prescribed by the participant's health care providers and will receive a home-based light (mild) physical activity program that begins approximately within one week after discharge from the hospital with the physical activity program starting approximately within the first week post-discharge from the hospital.
  Interventions: Behavioral: Light Physical Activity 1
- Light Physical Activity 2 (Experimental): Conventional treatment for cancer as prescribed by the participant's health care providers and will receive a home-based light (mild) physical activity program that begins approximately within one week after discharge from the hospital with the physical activity program starting approximately 7 weeks post-discharge from the hospital.
  Interventions: Behavioral: Light Physical Activity 2
- Support Education Activity (Active Comparator): Conventional treatment for cancer as prescribed by the participant's health care providers and will participate in a supportive cancer-related education activity each week for 6-weeks after returning home from the hospital.
  Interventions: Behavioral: Support Education Activity

INTERVENTIONS:
Behavioral: Light Physical Activity 1 — Light (mild) physical activity program that corresponds with normal every day activities of daily living (< 3.0 metabolic equivalents, METs), with a time commitment starting at 5 minutes a day 5 days a week gradually increasing to 30 minutes a day 5 days a week as you are able by week 6 as guided by your Registered Nurse researcher.
  The program begins approximately within one week after discharge from the hospital with the physical activity program starting approximately within the first week post-discharge from the hospital.
  Arms: Light Physical Activity 1
Behavioral: Light Physical Activity 2 — Light (mild) physical activity program that corresponds with normal every day activities of daily living (< 3.0 metabolic equivalents, METs), with a time commitment starting at 5 minutes a day 5 days a week gradually increasing to 30 minutes a day 5 days a week as you are able by week 6 as guided by your Registered Nurse researcher.
  The program begins approximately within one week after discharge from the hospital with the physical activity program starting approximately 7 weeks post-discharge from the hospital.
  Arms: Light Physical Activity 2
Behavioral: Support Education Activity — Participate in a supportive cancer-related education activity including a direct 10 - 15 minute phone conversation with a Registered Nurse researcher each week for 6-weeks after returning home from the hospital. Wear a pedometer each day of the study.
  Recording pedometer steps in the daily diary each day.
  Arms: Support Education Activity

SUMMARY:
Among 13 core symptoms across 3,106 breast, colorectal, prostate, and lung cancer patients, persons with lung cancer were the most symptomatic, with moderate to severe fatigue being reported with the greatest prevalence. This is a proposed randomized controlled trial of a novel rehabilitative intervention for persons with non-small cell lung cancer after surgery that promotes self-management of cancer-related fatigue (CRF) and is practical, portable, low cost, and safe. The results of the study will provide a novel exercise intervention, and its optimal timing, that helps a vulnerable population by reducing CRF severity and fatigability and is applicable to nearly all post-thoracotomy lung cancer patients.

DETAILED DESCRIPTION:
Persons with non-small cell lung cancer (NSCLC) report significantly more unmet supportive care needs than other cancer populations, yet they are among the most vulnerable and least studied. Two of the most prevalent unmet supportive care needs include overcoming fatigue and attaining adequate exercise to meet physical demands of daily living. Cancer-related fatigue (CRF) is a prevalent, persistent, and distressing symptom in the NSCLC population. Cancer-related fatigue correlates with greater severity of 15 other symptoms, leading to lower physical function for persons with NSCLC. Among 13 core symptoms across 3,106 breast, colorectal, prostate, and lung cancer patients, persons with lung cancer were the most symptomatic, with moderate to severe fatigue being reported with the greatest prevalence. While surgery is the standard curative treatment for NSCLC, no formal guidelines exist for post-surgical rehabilitation. This is a proposed randomized controlled trial (RCT) of a novel rehabilitative intervention for persons with NSCLC after surgery. The intervention promotes self-management of CRF and tests the intervention's impact on CRF severity and fatigability with analysis by age. Preliminary data included a two-arm RCT (R21 CA164515) incorporating the proposed intervention, where study goals were exceeded for recruitment (66%), retention (97%), adherence (93%), and acceptability. The 6-wk exercise intervention demonstrated preliminary efficacy in significantly reducing CRF severity and fatigability as compared to usual care, with mean CRF levels restored to levels lower than pre-surgery. The exercise group's functional performance exceeded usual care. No adverse events were reported; participants had a mean age of 67 with a mean of 8 comorbid conditions. The investigator's long-term goal is to develop interventions to increase perceived self-efficacy for CRF self-management in order to improve CRF, symptom status, functional status, and quality of life (QOL) for persons with NSCLC. The objective in this application is to determine the efficacy, optimal timing, and sustainability of this innovative home-based exercise intervention. This study has the potential to transform the current standard by providing a rehabilitative exercise intervention after surgery. The intervention is home-based, self-paced, and builds in duration upon discharge from the hospital after surgery. Aim 1: Determine efficacy by comparing the immediate intervention group with wait-list control (usual care) and attention control by age. Aim 2: Determine efficacy of initiating the exercise intervention 6 wks post-discharge and compare results with the immediate intervention group for all ages. Aim 3: Determine the immediate intervention's sustainability by analyzing 3a) rates of extension, adherence, and retention; 3b) acceptability; and 3c) efficacy of primary and secondary outcomes. IMPACT: The results of this study will provide a novel exercise intervention, and its optimal timing, and fill the gap for a vulnerable population by providing a practical, portable, and low-cost means of reducing CRF severity and fatigability that is enjoyable and applicable to nearly all post-thoracotomy lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* At least 18 years of age (Michigan) and 19 years of age in (Nebraska)
* With suspected non-small cell lung cancer to be confirmed after surgery
* Karnofsky Performance Status score of at least 70%
* Thoracic surgeon approval pre- and post-surgery
* Medically stable comorbid conditions allowing for non-small cell lung cancer surgery clearance
* Has phone access capability
* Able to speak and write English
* Able to hear and speak for phone interviews
* Owns a television
* Lives within 2 hours driving distance of recruitment site

Exclusion Criteria:

* Severe impairment of sight, hearing, speaking
* Active treatment for malignancy within past 3 months (other than non-melanoma skin cancer or long-term hormonal treatment for common cancers such as breast and prostate if disease is stable
* Weight greater than 330 pounds
* History of photosensitive seizures
* Any condition or disorder that would impede safe participation as directed
* Plans to relocate outside the area during the study period or unable to fully participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Cancer-Related Fatigue Severity as assessed using an 11-point rating scale | about 6 weeks after discharge from the hospital
  Degree of cancer-related fatigue severity on an 11-point scale (0-10, 10 = most severe)
Cancer-Related Fatigue Fatigability as assessed using the 6 minute walk test | about 6 weeks after discharge from the hospital
  Average fatigue level while performing the 6 minute walk test on an 11-point scale (0-10, 10 = most severe)

SECONDARY OUTCOMES:
Other Symptoms Severity | about 6 weeks after discharge from the hospital
  Severity of multiple symptoms and symptoms interference on daily life on an 11-point scale (0-10, 10 = most severe and most interference)
Perceived Self-Efficacy for Fatigue Self-Management | about 6 weeks after discharge from the hospital
  A persons's perception of ability to manage fatigue on an 11-point scale (0-10, 10 = very certain)
Self-Efficacy for Walking Duration | about 6 weeks after discharge from the hospital
  A person's perception to complete incremental 5-minute periods of walking using an 11-point scale (0-100%, 100% = very confident)
Activities-Specific Balance Confidence | about 6 weeks after discharge from the hospital
  A person's perception of balance during every day activities using an 11-point scale (0-100%, 100% = very confident
Steps Per Day | about 6 weeks after discharge from the hospital
  Performance in average number of walking steps taken per day per week
Functional Status Performance | about 6 weeks after discharge from the hospital
  Performance of daily mental and physical activities that people do in the normal course of their lives measured with eight subscales that focus on the physical and mental health components producing normative scores (0-100, 100 = higher functional status)
Quality of Life as assessed using a 6-point rating scale | about 6 weeks after discharge from the hospital
  Satisfaction with various aspects of life and the importance of each aspect of life to the person using a 6 point-rating scale (1-6, 6 = very satisfied and very important)

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Hoffman, PhD, RN, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
We will disseminate the results from this study at national/international meetings. We also expect that the findings of this study will be disseminated through scientific journals with multiple manuscripts prepared by the investigators from this study for publication in peer-reviewed journals. The investigators agree to continue to abide by the NIH Public Access Policy by submitting final peer-reviewed journal manuscripts to the digital archive, PubMed Central, upon acceptance for publication.